CLINICAL TRIAL: NCT03254303
Title: Intravenous Cannulation In Children During Sevoflurane Induction: Which Time is Adequate
Brief Title: Intravenous Cannulation In Children During Sevoflurane Induction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leila mansali stambouli (Other)
Responsible Party: Sponsor-Investigator, Leila mansali stambouli, Principal Investigator and Clinical Professor, University of Monastir
Organization: University of Monastir (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: OMB: 0925-0586
Record Dates: First submitted 2017-08-11; First posted 2017-08-18 (Actual); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Catheterization
Keywords: Sevoflurane, Catheterization, Anesthetics Inhalation, child
MeSH Terms: interventions — Population Groups

STUDY DESIGN:
Intervention Model Description: randomized and crossover assignemnt
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: particippant, investigator, outcomes assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 60s (group E) (Other): The Time of catheterization at 60s (group E) was applied in this study group,after sevoflurane inhalation induction, 30 children have a catheterization after a time of 60 seconds following the eye closure and the loss of lid reflex.Difficulty with intravenous catheterization, limb movement and laryngospasm were recorded.Difficulty of catheterization in group 60 s
  Interventions: Other: Difficulty of catheterization in group 60 s
- 90s (groupe L) (Other): In this study group,after sevoflurane inhalation induction, 30 children have a catheterization after a time of 90 seconds following the eye closure and the loss of lid reflex.Difficulty with intravenous catheterization, limb movement and laryngospasm were recorded.Difficulty of catheterization in group 90 s
  Interventions: Other: Difficulty of catheterization in group 90 s
- 120s (groupe L) (Other): In this study group,after sevoflurane inhalation induction, 30 children have a catheterization after a time of 120 seconds following the eye closure and the loss of lid reflex.Difficulty with intravenous catheterization, limb movement and laryngospasm were recorded.Difficulty of catheterization in group 120 s
  Interventions: Other: Difficulty of catheterization in group 120 s

INTERVENTIONS:
Other: Difficulty of catheterization in group 60 s
  Arms: 60s (group E)
Other: Difficulty of catheterization in group 90 s
  Arms: 90s (groupe L)
Other: Difficulty of catheterization in group 120 s
  Arms: 120s (groupe L)

SUMMARY:
This interventional simple-blind,randomized trial has included 90 children of American Society of Anesthesiologist (ASA) physical status I or II aged between 1 to 12 years of either sex, scheduled for for outpatient minor surgery under general anesthesia. This study examined whether one should make iv attempts during the early induction period (at 60 seconds) or lately (90 or 120 s) and waiting until the child receives additional sevoflurane inhalation anesthesia.

DETAILED DESCRIPTION:
We conducted a prospective randomized study, after obtaining Institutional review board approval, which didn't require written parental consent. Children age 1-12 years, undergoing elective general anesthesia via an inhalation induction were randomized to one of three groups of 30 patients each one, for iv placement, either 60s (group E), 90 or 120 s (group L) following loss of lid reflex. Movement on iv placement and incidence of laryngospasm were determined. Difficulty with iv placement was also recorded. Statistical analysis included contingency testing, ANOVA, and non parametric testing. A P-value <0.05 was considered significant.

ELIGIBILITY:
Inclusion Criteria:

* children with American Society of Anesthesiologist (ASA) physical status I or II
* age between 1 and 12 years of either sex,
* were scheduled for outpatient minor surgery under general anesthesia

Exclusion Criteria:

* age <1 and >12 years
* patients with full stomach
* a history of gastric reflux
* history of convulsions, cardiovascular or neuromuscular disease
* suspected difficult airway and hyper-reactive airway disease

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2016-10-31 (Actual); Study Completion 2016-10-31 (Actual)

PRIMARY OUTCOMES:
Success of intravenous insertion | from the end of study period of time after the loss of eyelash reflex to successful cannulation less than 30 seconds
  success insertion of intravenous cannula was achieved at the first attempt less than 30 seconds

SECONDARY OUTCOMES:
limb movement | from the end of study period of time after the loss of eyelash reflex to successful cannulation less than 30 seconds
  The movement was classified using the scale:
  (0 No movement, 1 movement) The incidence of laryngospasm was defined as the sudden complete or partial loss of air exchange with concurrent loss of a capnographic wave.
  The movement was classified using the scale:
  (0 No movement, 1 movement) The incidence of laryngospasm was defined as the sudden complete or partial loss of air exchange with concurrent loss of a capnographic wave.
  • The movement was classified using the scale: (0 No movement, 1 movement)
  • The movement was classified using the scale: (0 No movement, 1 movement) The limb movement was classified using the scale:0 No movement, 1 movement)

OTHER OUTCOMES:
laryngospasm | from the end of study period of time after the loss of eyelash reflex to successful cannulation less than 30 seconds
  laryngospasm was defined as the sudden complete or partial loss of air exchange with concurrent loss of a capnographic wave.

CONTACTS AND LOCATIONS:
Overall Officials: leila Mansali Stambouli, MD PhD, Principal Investigator — University Hospital of Fattouma Bourguiba Monastir TUNISIA

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Choudhry DK, Stayer SA, Schwartz RE, Pasquariello CA. Early intravenous cannulation in children during inhalational induction of anaesthesia. Paediatr Anaesth. 1998;8(2):123-6. doi: 10.1046/j.1460-9592.1998.00731.x. PMID 9549737
- [Result] Schwartz D, Connelly NR, Gutta S, Freeman K, Gibson C. Early intravenous cannulation in children during sevoflurane induction. Paediatr Anaesth. 2004 Oct;14(10):820-4. doi: 10.1111/j.1460-9592.2004.01315.x. PMID 15385009